CLINICAL TRIAL: NCT03949400
Title: Effects of Exercise Therapy and Soft Brace on Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: FOU-UU-2018-007
Record Dates: First submitted 2018-10-02; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-02

CONDITIONS: Rehabilitation; Treatment Outcome; Pain; Knee Brace; Outcome Assessment (Health Care); Recovery of Function; Patient Reported Outcome Measures; Adults; Osteoarthritis, Knee
MeSH Terms: conditions — Pain; Osteoarthritis, Knee | interventions — Exercise Therapy; Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with knee OA: Patients diagnosed with knee OA and assigned to undergo exercise therapy and education.
  Interventions: Other: Exercise therapy and education.

INTERVENTIONS:
Other: Exercise therapy and education. — Exercise therapy and education, physiotherapy rehab at Aalborg Municipality

SUMMARY:
The primary aim of the study is to investigate the effects of supervised exercise therapy and education on the immediate response to using a soft knee brace in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
Study type: observational Estimated enrollment: 40 participants Observational model: cohort Time perspective: prospective

Inclusion Criteria:

Assigned for exercise and education due to knee osteoarthrosis Age 18 years or older at the time of recruitment Able to read and understand Danish

Exclusion Criteria:

Not mentally able to reply to the questionnaire

Patients are tested with and without the brace before starting the exercise therapy and education program and re-tested with and without the brace after completing the treatment program (6 weeks) and again at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Assigned for exercise and education due to knee osteoarthrosis Age 18 years or older at the time of recruitment Able to read and understand Danish

Exclusion Criteria:

Not mentally able to reply to the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with knee OA and assigned to undergo exercise therapy and education
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-04-24 (Estimated); Study Completion 2029-05-20 (Estimated)

PRIMARY OUTCOMES:
Pain - Numerical rating scale (NRS) | 6+12 weeks follow-up
  NRS is the most common pain scale for quantification pain. The respondent selects a whole number on a scale from 0-10, that best reflects the intensity of his/her pain. 0 being no pain, 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Y-balance test (YBT) | 6+12 weeks follow-up
  The YBT test is a test commonly used in clinical practice to investigate functional balance. The YBT is based on the Star Excursion Balance Test and it has been thoroughly researched. Measured with and without the soft knee brace at baseline, after the treatment program and at 12weeks.
Self-perceived knee stability question | 6+12 weeks follow-up
  Self-reported by the patients.
40-meter walk test | 6+12 weeks follow-up
  A test of walking speed over shirt distances and changing direction during walking

OTHER OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) (continous) | 6+12 weeks follow-up
  An instrument to assess the patient's opinion about their knee and associated problems. KOOS has been evaluated and compared to other instruments in several studies. Measured at baseline, after the treatment program and at 12weeks.
Pain manikin | 6+12 weeks follow up
  Self-reported pain assessment by the patients.
Likert scale | 6+12 weeks follow-up
  Self-reported by the patients
Analgetic pain medication intake | 6+12 weeks follow-up
  Self-reported by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachmann, Study Director — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- Aalborg Municipality, training unit west, Aalborg, Nothern, Denmark

IPD SHARING:
Plan to Share IPD: Undecided